CLINICAL TRIAL: NCT03354156
Title: Effect of Statins on Epigenetic Reprogramming of Monocytes in Patients With Elevated Levels of LDL
Brief Title: The Effect of Statin Treatment on Trained Innate Immunity
Acronym: SIMPEL
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: AIDS Malignancy Consortium (Network); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL50608.091.14
Record Dates: First submitted 2016-04-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2016-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * plasma
  * chromatin and RNA from monocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High-LDL: patients with LDL cholesterol levels of >4.9 mmo/l, who have not been treated with statins in the past years, and who have an indication for treatment with statins.
  Interventions: Drug: statin treatment
- Control: control subjects with an LDL cholesterol level of <3.5 mmol/l

INTERVENTIONS:
Drug: statin treatment — The patients with elevated LDL receive statin treatment in the context of normal patient care (so this is NOT an intervention of the study)
  Groups: High-LDL

SUMMARY:
The innate immune system plays a pivotal role in the development and progression of atherosclerosis. Recently, it was reported that monocytes can develop a long-lasting immunological memory after stimulation with various microorganisms, which has been termed 'trained innate immunity'. This memory is induced by epigenetic reprogramming, in particular trimethylation of lysine 4 at histone 3 (H3K4me3).

In this study, the investigators aim to investigate the immunophenotype of circulating monocytes in patients with elevated LDL cholesterol levels and the effect of statins on this phenotype.

DETAILED DESCRIPTION:
The innate immune system plays a pivotal role in the development and progression of atherosclerosis. Recently, it was reported that monocytes can develop a long-lasting immunological memory after stimulation with various microorganisms, which has been termed 'trained innate immunity'. This memory is induced by epigenetic reprogramming, in particular trimethylation of lysine 4 at histone 3 (H3K4me3).

The main objective is to study whether circulating monocytes of patients with elevated levels of LDL have a phenotype of trained innate immunity compared to control patients. Subsequently the investigators will study the effect of treatment with statins on the increased inflammatory response and epigenetic changes of the innate immune system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Elevated LDL levels (>4.9 mmol/l)
* Decision made by treating physician to initiate statin treatment

Exclusion Criteria:

* previous cardiovascular events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the outpatient clinics of the Radboudumc, AMC, or Erasmus MC, with LDL cholesterol levels >4.9 mmol/l, who will treated with statins according to current guidelines, will be will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cytokine production capacity | baseline
  Cytokine production capacity of PBMC's at baseline in patients with elevated and normal cholesterol levels

SECONDARY OUTCOMES:
Cytokine production capacity | Three months after start of statin treatment
  Cytokine production capacity of PBMC's at baseline in patients with elevated and normal cholesterol levels
Epigenetic modifications in the promoter regions of the pro-inflammatory cytokines in monocytes. | baseline
  Epigenetic modifications in the promoter regions of the pro-inflammatory cytokines in monocytes.
Epigenetic modifications in the promoter regions of the pro-inflammatory cytokines in monocytes. | Three months after start of statin treatment
  Epigenetic modifications in the promoter regions of the pro-inflammatory cytokines in monocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No